[On local headed notepaper]

## ObservAtional study to investigate Surgical site Infection in ulcerated Skin cancers (OASIS):

Observational study to estimate the proportion of post-operative infection following excision of ulcerated skin tumours.

| Sponsor: | Cardiff and Vale University Health Board (CAVUHB) |
|--------------|---------------------------------------------------|
| Sponsor ref: | RD 17/DEC/7165 |
| | UK Dermatology Clinical Trials Network (UK DCTN) |
| Funders: | Dermatology Forum for Wales |
| | CAVUHB Dermatology Department Research Funds |
| Funder ref: | UK DCTN Pump Priming Award 2017 |
| REC ref: | 19/SC/0047 |
| IRAS number: | 243011 |
| NCT number: | NCT03782727 |

| Participant ID: |
|-----------------|

## OASIS Observational Prospective Study

## Please initial

| | PARTICIPANT CONSENT FORM | each box |
|---|---|---|
| 1. | I confirm that I have read and understood the information sheet (version 1.5, date 18/09/19) for the above study. I have had the opportunity to ask questions and these have been answered satisfactorily. | |
| 2. | I understand that my participation in this study is voluntary and that I am free to withdraw at any time without my medical care or legal rights being affected. I understand that if I withdraw then none of my data, including wound photographs will be included in the results of the study. I understand that I cannot withdraw data after it has been anonymised for analysis. | |
| 3. | I understand that relevant sections of my healthcare records and data collected during the study may be looked at by individuals from the research team, the regulatory authorities, [Oxford University Hospital NHS Foundation Trust/University Hospitals Birmingham NHS Foundation Trust] or Cardiff & Vale Health Board overseeing the research in order to check that the study is being carried out correctly. I give permission for these individuals to have access to the relevant parts of my medical records. | |
| 4. | I understand that the clinical/research team will keep secure records at the hospital and in Cardiff University Centre for Trials Research (including name, address/ e-mail address and phone number) which will allow me to be followed up by questionnaire four weeks after surgery and provide 'wound selfies'. | |
| 5. | I consent to the secure storage in compliance with Data Protection requirements, including paper and electronic, of personal information for the purposes of this study, until five years after the end of the study when these details will be destroyed. | |
| 6. | I agree to allow any information (including photos –'wound selfies') or results arising from this study to be used for healthcare and/or further medical research upon the understanding that my identity will remain anonymous. | |
| 7. | I agree to having a swab taken of the ulcerated skin cancer (Cardiff and Vale UHB participants) | |

| 8. I agree to take par | t in the study | |
|-------------------------------|----------------|-----------|
| Name of Participant | Date | Signature |
| Name of Person taking consent | Date | Signature |